CLINICAL TRIAL: NCT07254923
Title: Three Brief Psychological Interventions for Acute Pain in Inpatients in Boyacá: Randomized Three-Arm Clinical Trial
Brief Title: Three Brief Psychological Interventions for Acute Pain in Inpatients in Boyacá
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pedagógica y Tecnológica de Colombia (Other)
Collaborators: ESE Hospital Regional de Sogamoso (Unknown); ESE Hospital Santa Marta de Samacá (Unknown); ESE Santiago de Tunja (Unknown); ESE Hospital Regional de Chiquinquirá (Unknown)
Responsible Party: Principal Investigator, Andrés Felipe Calvo-Abaunza, Full-Time Lecturer, School of Psychology, Universidad Pedagógica y Tecnológica de Colombia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT-PSI-01
Record Dates: First submitted 2025-11-14; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pain Management; Pain Acute
Keywords: body scanning; ABC; Guided Imagery; Breathing Exercises; Acute Pain; Pain Measurement; Pain Management; Inpatients; Randomized Controlled Trial
MeSH Terms: conditions — Agnosia; Acute Pain | interventions — Imagery, Psychotherapy; Osteogenesis, Distraction; Whole Body Imaging

STUDY DESIGN:
Intervention Model Description: Individually randomized, three-arm, parallel assignment (1:1:1) comparing two brief behavioral techniques-body-scan mindfulness and guided imagery/distraction-with an active comparator (CBT-based psychoeducation). Randomization uses computer-generated variable block sizes with allocation concealment until assignment. Open-label, single-session interventions delivered at the bedside with pre- and post-session pain assessment.
Who Masked: Outcomes Assessor
Masking Description: Single-blind (outcomes assessor). An external evaluator, not present during the intervention and unaware of group assignment (arms labeled A/B/C), administers and scores prespecified secondary outcomes-Pain Self-Efficacy Questionnaire (PSEQ-10), Pain Catastrophizing Scale (PCS), and Hospital Anxiety (HADS-A)-and has no access to baseline scores at the time of assessment. Participants and interventionists are not blinded. The primary outcome (acute pain 0-10) is patient-reported at bedside. Allocation is concealed until assignment (computer-generated variable blocks). Any inadvertent unblinding is documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guided Imagery (B) (Experimental): Single, bedside session (~15-20 min) of therapist-guided guided imagery that redirects attention from pain toward neutral or pleasant sensory images and simple attentional shifts. Delivered seated or semi-reclined in addition to usual care. Pain is rated immediately before and after the session (0-10). A protocolized slow deep-breathing rescue (≤5 min) may be offered if pain remains very high or the technique cannot be completed.
  Interventions: Behavioral: Guided Imagery
- Body-Scan Mindfulness (A) (Experimental): Single, bedside body-scan mindfulness session (~12-20 min) guiding non-judgmental attention sequentially through body areas, including sites without pain, to foster an open, accepting stance toward the pain experience. Delivered seated or semi-reclined with usual care continuing. Pain is rated immediately before and after (0-10). Rescue slow deep-breathing (≤5 min) may be used if needed.
  Interventions: Behavioral: Body-Scan Mindfulness
- CBT-Based Psychoeducation (ABC Model) (C) (Active Comparator): Brief, structured explanation of the ABC cognitive-behavioral model applied to pain (~10-15 min) using a practical example; no skills training or practice. Serves as an active comparator controlling for time and attention. After the immediate post-session pain assessment, participants in this arm receive one of the two techniques (body-scan mindfulness or guided imagery) during the same visit (equity measure). Rescue slow deep-breathing (≤5 min) available per protocol.
  Interventions: Behavioral: CBT-Based Psychoeducation (ABC Model)

INTERVENTIONS:
Behavioral: Guided Imagery — Single, bedside session (~15-20 minutes) of therapist-guided guided imagery/distraction that redirects attention from pain toward neutral or pleasant sensory images and simple attentional shifts. Seated or semi-reclined, conversational and supportive, in addition to usual care. Pain is rated immediately before and after the session (0-10).
  Other Names: Distraction
  Arms: Guided Imagery (B)
Behavioral: Body-Scan Mindfulness — Single, bedside body-scan mindfulness session (~12-20 minutes) guiding non-judgmental attention sequentially through body areas-including regions without pain-to cultivate an open, accepting stance toward pain. Delivered seated or semi-reclined with usual care continuing. Pain is rated immediately before and after (0-10).
  Other Names: body scan
  Arms: Body-Scan Mindfulness (A)
Behavioral: CBT-Based Psychoeducation (ABC Model) — Brief, structured explanation of the ABC cognitive-behavioral model (thoughts-emotions-behaviors) applied to pain (~10-15 minutes) using a practical example; no skills training or practice. Serves as an active comparator controlling for time and attention. After the immediate post-session pain assessment, participants in this arm receive one of the two techniques (body-scan mindfulness or guided imagery) during the same visit (equity measure).
  Other Names: ABC Model Education; Cognitive Behavioral Psychoeducation
  Arms: CBT-Based Psychoeducation (ABC Model) (C)

SUMMARY:
This study evaluates two brief, non-drug psychological techniques-body-scan mindfulness and guided imagery/distraction-delivered as a single bedside session to reduce acute pain in adults admitted to short-stay inpatient wards or emergency observation units in Boyacá, Colombia. Participants are randomly assigned (1:1:1) to body-scan mindfulness, guided imagery/distraction, or a brief cognitive-behavioral psychoeducation session (active comparator). Each session lasts under 20 minutes and usual medical care continues. Pain intensity (0-10) is recorded within 5 minutes before the session and within 2 minutes after completion on the same day. If pain remains very high (e.g., ≥8-9/10) or the activity cannot be completed, up to 5 minutes of supervised slow deep-breathing may be offered as rescue, and the clinical team may adjust analgesics per routine care. Secondary measures (specified in Outcome Measures) include patient satisfaction, feasibility (session duration and completion), use of rescue measure, and adverse events; exploratory data may include short-term psychological scales collected by a blinded assessor and the association with length of stay during the current admission. Adults aged ≥18 years with acute pain ≤7 days and baseline pain ≥4/10 may be eligible. The study takes place across four public hospitals in Boyacá, Colombia.

DETAILED DESCRIPTION:
This is a parallel-group, open-label, three-arm randomized trial (1:1:1) in short-stay inpatient wards and emergency observation units at four public hospitals in Boyacá, Colombia. The objective is to estimate the immediate effect of a single, brief bedside behavioral session on acute pain while routine medical care continues unchanged. Clinically stable adults provide written informed consent prior to any study procedures.

Participants are randomized to one of three groups. Group A (body-scan mindfulness) receives a guided practice that cultivates open, non-judgmental attention across body regions, including areas without pain, to modulate the nociceptive experience. Group B (guided imagery/distraction) receives a session using neutral/pleasant imagery and simple attentional shifts intended to redirect focus away from painful sensations. Group C (CBT-based psychoeducation; ABC model) serves as an active comparator and consists of a brief, structured explanation of the relationship between thoughts, emotions, and sensations using a practical example; no skills training is included. Each technique is delivered once (<20 minutes) by trained study personnel (e.g., psychology staff). The attending clinical team (physicians/nurses) is informed of participation and may adjust routine care as needed, but does not deliver study techniques or collect study outcomes. If post-session pain remains very high or a participant cannot complete the assigned activity, up to 5 minutes of supervised slow deep-breathing may be offered as a rescue measure; any analgesic adjustments are per routine care and are not protocol-driven.

Randomization uses a computer-generated sequence with variable permuted block sizes (1:1:1) prepared in advance and stored in a password-protected spreadsheet with locked sheets/cells and restricted access. Assignment is centralized: after eligibility confirmation, informed consent, and documentation of baseline pain, the enrolling clinician contacts the study coordinators, who control the file and release the next sequential assignment. Block sizes and the remaining sequence are concealed from enrolling staff; each release is time-stamped and logged to preserve allocation concealment and balanced assignment across arms.

Assessments follow standardized procedures. The primary endpoint is the immediate pre- to post-session change in pain intensity; operational details (instruments and exact time windows) are specified in Outcome Measures and captured on case-report forms. Where feasible, a blinded outcomes assessor administers only the post-session psychological scales 5-10 minutes after the session (e.g., PSEQ-10, PCS, HADS-A) and has no access to pain ratings or allocation files. Pain ratings and the participant satisfaction questionnaire are recorded at bedside by study personnel involved in the session. The pre-session length of stay during the index admission may also be abstracted from the medical record as specified in Outcome Measures.

The analysis overview is prespecified. The primary comparison of immediate pain change across arms will use a linear model under intention-to-treat, with post-session pain as the dependent variable and baseline pain and study site as covariates; adjusted mean differences with 95% confidence intervals will be reported. Secondary endpoints (e.g., safety and patient-reported satisfaction) will be summarized with models appropriate to their scale. Exploratory analyses will compare post-session psychological scale scores across arms and examine the association between pre-session length of stay and pain change. Missing post-session pain data are expected to be minimal; if present, prespecified sensitivity analyses (e.g., complete-case vs simple imputation) will be conducted. No multiplicity adjustment is planned for secondary/exploratory outcomes. Ethics approvals were obtained from the participating institutions; written informed consent is required prior to any study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Admitted to short-stay inpatient or emergency observation units at participating hospitals (same index admission).
* Acute pain ≤7 days with baseline pain ≥4/10 on a 0-10 numeric/visual scale.
* Clinically stable and able to remain at bedside for ~30-40 minutes (consent, baseline, single session, post-session assessment).
* Analgesic regimen stable ≥1 hour before baseline pain rating (no planned change during the ~20-minute study window unless clinically required).
* Able to understand simple instructions and communicate pain ratings (verbal or pointing) and to provide written informed consent.

Exclusion Criteria:

* Cancer-related pain or chronic pain >6 months (e.g., widespread musculoskeletal pain/fibromyalgia).
* Active inflammatory/degenerative rheumatic disease causing ongoing daily pain that would confound acute pain ratings (e.g., rheumatoid arthritis flare, advanced osteoarthritis, severe osteoporosis-related pain).
* Cognitive impairment/dementia, delirium, or acute severe psychiatric disturbance that prevents consent or reliable self-report.
* Respiratory conditions that contraindicate slow deep-breathing rescue (e.g., decompensated COPD, acute asthma, need for high-flow oxygen or ventilatory support).
* Hemodynamic or clinical instability (e.g., need for urgent procedure; in resuscitation/reanimation area; RASS ≤ -3; MAP <65 mmHg or SBP <90 mmHg; SpO₂ <90% despite usual oxygen) at screening.
* Participation in another interventional study targeting pain during the same admission.
* Refusal to participate or withdrawal of consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-16 (Estimated)

PRIMARY OUTCOMES:
Change in acute pain intensity (0-10 Pain Thermometer) from pre- to post-session | Two assessments on the same calendar day: ≤5 minutes before session start and ≤2 minutes after session end.
  Patient-reported Pain Thermometer adapted from VAS/NRS; 0 = no pain, 10 = worst imaginable pain. Higher scores indicate more pain. Change score = post-session minus pre-session (negative values indicate pain reduction).

SECONDARY OUTCOMES:
Patient satisfaction with the session | One assessment ≤5 minutes after session end (same calendar day).
  Brief satisfaction questionnaire (two Likert items 1-10; higher scores = greater satisfaction). Open comments are collected but not scored. Report the mean satisfaction score (1-10).
Participants requiring protocolized rescue slow deep-breathing | From session start until ≤10 minutes after session end (same calendar day).
  Per protocol, up to 5 minutes of slow deep-breathing is offered if post-session pain is very high (e.g., ≥8/10) or the technique cannot be completed. Report the proportion of participants for whom rescue was used (Yes/No).
Pain Self-Efficacy (PSEQ-10) - change from pre- to post-session | One assessment 5-10 minutes after session end (same calendar day).
  PSEQ-10 (10 items, 0-6 each; total 0-60). Higher scores = greater pain self-efficacy. Administered and scored by a blinded outcomes assessor. Report change score (post minus pre).
Pain Catastrophizing (PCS) - change from pre- to post-session | One assessment 5-10 minutes after session end (same calendar day).
  Pain Catastrophizing Scale (PCS; 13 items, 0-4 per item; total 0-52). Subscales: Rumination, Magnification, Helplessness. Higher scores indicate greater catastrophizing. Administered and scored by a blinded outcomes assessor at a single post-session time point; intended to characterize cognitive-affective responses to pain during the index admission.
Hospital Anxiety (HADS-A) - change from pre-session to post-session | One assessment 5-10 minutes after session end (same calendar day).
  7-item Hospital Anxiety subscale (0-21). Higher scores = more anxiety. Administered by a blinded outcomes assessor.

OTHER OUTCOMES:
Days hospitalized immediately before the session (pre-session length of stay) | Calculated on the day of the intervention, from index hospital admission/observation start to session start for the same hospitalization; assessed for admissions up to 30 days prior to the session.
  Continuous days calculated as (session start - admission/observation start) ÷ 24 hours; same-day = 0.0 days; transfers use arrival to index hospital. Recorded to explore whether pre-session stay moderates the change in pain; it is not expected to be altered by the single session.

CONTACTS AND LOCATIONS:
Locations (4):
- Colombia (4):
  - ESE Hospital Regional de Chiquinquirá, Chiquinquirá, Departamento de Boyacá
  - ESE Hospital Santa Marta de Samacá, Samacá, Departamento de Boyacá
  - ESE Hospital Regional de Sogamoso, Sogamoso, Departamento de Boyacá
  - ESE Santiago de Tunja, Tunja, Departamento de Boyacá

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary outcome will be shared. Direct identifiers will be removed and indirect identifiers minimized in accordance with Colombian data protection law and IRB approvals.
Supporting Information: Study Protocol, ICF
Time Frame: Within 12 months after publication of the primary results; available for 24 months thereafter.
Access Criteria: Available upon reasonable request to the corresponding author/UPTC data custodian for qualified researchers with a methodologically sound proposal and ethics approval, after signing a Data Use Agreement.

REFERENCES:
- [Background] Sun JN, Chen W, Zhang Y, Zhang Y, Feng S, Chen XY. Does cognitive behavioral education reduce pain and improve joint function in patients after total knee arthroplasty? A randomized controlled trial. Int Orthop. 2020 Oct;44(10):2027-2035. doi: 10.1007/s00264-020-04767-8. Epub 2020 Aug 8. PMID 32772319
- [Background] Miller-Matero LR, Coleman JP, Smith-Mason CE, Moore DA, Marszalek D, Ahmedani BK. A Brief Mindfulness Intervention for Medically Hospitalized Patients with Acute Pain: A Pilot Randomized Clinical Trial. Pain Med. 2019 Nov 1;20(11):2149-2154. doi: 10.1093/pm/pnz082. PMID 31329961
- [Background] Maniaci G, Daino M, Iapichino M, Giammanco A, Taormina C, Bonura G, Sardella Z, Carolla G, Cammareri P, Sberna E, Clesi MF, Ferraro L, Gambino CM, Ciaccio M, Rispoli L, La Cascia C, La Barbera D, Quattrone D. Neurobiological and Anti-Inflammatory Effects of a Deep Diaphragmatic Breathing Technique Based on Neofunctional Psychotherapy: A Pilot RCT. Stress Health. 2024 Dec;40(6):e3503. doi: 10.1002/smi.3503. Epub 2024 Nov 14. PMID 39543797
- [Background] Joseph AE, Moman RN, Barman RA, Kleppel DJ, Eberhart ND, Gerberi DJ, Murad MH, Hooten WM. Effects of Slow Deep Breathing on Acute Clinical Pain in Adults: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Evid Based Integr Med. 2022 Jan-Dec;27:2515690X221078006. doi: 10.1177/2515690X221078006. PMID 35225720
- [Background] Jafari H, Gholamrezaei A, Franssen M, Van Oudenhove L, Aziz Q, Van den Bergh O, Vlaeyen JWS, Van Diest I. Can Slow Deep Breathing Reduce Pain? An Experimental Study Exploring Mechanisms. J Pain. 2020 Sep-Oct;21(9-10):1018-1030. doi: 10.1016/j.jpain.2019.12.010. Epub 2020 Jan 22. PMID 31978501
- [Background] Hanley AW, Gililland J, Garland EL. To be mindful of the breath or pain: Comparing two brief preoperative mindfulness techniques for total joint arthroplasty patients. J Consult Clin Psychol. 2021 Jul;89(7):590-600. doi: 10.1037/ccp0000657. Epub 2021 Jun 24. PMID 34165999
- [Background] Garcia-Galicia A, Diaz-Diaz JF, Montiel-Jarquin AJ, Gonzalez-Lopez AM, Vazquez-Cruz E, Morales-Flores CF. Validity and consistency of an outpatient department user satisfaction rapid scale. Gac Med Mex. 2020;156(1):47-52. doi: 10.24875/GMM.19005144. PMID 32026871
- [Background] Ferrer-Pena R, Gil-Martinez A, Pardo-Montero J, Jimenez-Penick V, Gallego-Izquierdo T, La Touche R. Adaptation and validation of the Spanish version of the graded chronic pain scale. Reumatol Clin. 2016 May-Jun;12(3):130-8. doi: 10.1016/j.reuma.2015.07.004. Epub 2015 Aug 19. English, Spanish. PMID 26298083
- [Background] Dilek B, Ayhan C, Yagci G, Yakut Y. Effectiveness of the graded motor imagery to improve hand function in patients with distal radius fracture: A randomized controlled trial. J Hand Ther. 2018 Jan-Mar;31(1):2-9.e1. doi: 10.1016/j.jht.2017.09.004. Epub 2017 Nov 6. PMID 29122370
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Darnall BD, Abshire L, Courtney RE, Davin S. Upskilling pain relief after surgery: a scoping review of perioperative behavioral intervention efficacy and practical considerations for implementation. Reg Anesth Pain Med. 2025 Feb 5;50(2):93-101. doi: 10.1136/rapm-2024-105601. PMID 39909552
- [Background] Birch S, Stilling M, Mechlenburg I, Hansen TB. No effect of cognitive behavioral patient education for patients with pain catastrophizing before total knee arthroplasty: a randomized controlled trial. Acta Orthop. 2020 Feb;91(1):98-103. doi: 10.1080/17453674.2019.1694312. Epub 2019 Nov 25. PMID 31762342